CLINICAL TRIAL: NCT02406976
Title: Effect of Physical Exercise on Different Approaches to Treatment of Morbid Obesity
Brief Title: Effect Physical Exercise in Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0328
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Morbid Obesity
Keywords: Exercise; Morbidity Obesity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- G1- EXERCISE (Experimental): The group will Participate in an physical exercise program twice a week. This program consists of 20 minutes of aerobic exercises of low intensity (2-4 on the Borg scale) in the rhythm of different songs that encourage their implementation. After these exercises will be performed five minutes of stretching exercises.
  Interventions: Other: G1 -Exercise; Other: G3- Control
- G2- EXERCISE AND LIFESTYLE (Experimental): This groups will receive the same intervention of G1 group, associated with the weekly group with a psychologist.
  These groups worked techniques of cognitive behavioral therapy based on principles of learning, in order to promote and maintain new healthy behaviors, as well as the reduction or elimination of undesirable conduct.
  Interventions: Behavioral: G2- Exercise and Lifestyle; Other: G3- Control
- G3- CONTROL (Active Comparator): This group will keep the routine treatment in outpatient of bariatric surgery. This treatment consists of individual consultations and 05 (five) information meetings organized by the multidisciplinary team composed by the surgeon, endocrinologist, psychologist, psychiatrist, nutritionist, physical education teacher, pulmonologist, cardiologist and nurse. The G1 and G2 will also receive this intervention.
  Interventions: Other: G3- Control

INTERVENTIONS:
Other: G1 -Exercise — 20 minutes of aerobic exercises of low intensity (2-4 on the Borg scale) in the rhythm of different songs that encourage their implementation. After these exercises will be performed five minutes of stretching exercises.
  Furthermore the similar treatment to G3.
  Arms: G1- EXERCISE
Behavioral: G2- Exercise and Lifestyle — Exercise more techniques of cognitive behavioral therapy based on principles of learning, in order to promote and maintain new healthy behaviors and the reduction or elimination of undesirable conduct.
  Furthermore the similar treatment to G3.
  Arms: G2- EXERCISE AND LIFESTYLE
Other: G3- Control — Routine treatment in outpatient of bariatric surgery. Consists of individual consultations and 05 (five) information meetings organized by the multidisciplinary team composed by the surgeon, endocrinologist, psychologist, psychiatrist, nutritionist, physical education teacher, pulmonologist, cardiologist and nurse. The G1 and G2 will also receive this intervention.

SUMMARY:
This objective study to verify the effect of physical training with and without behavioral cognitive therapy, compared with controls, in functional capacity and cardio-metabolic profile in individuals with morbidly obese

DETAILED DESCRIPTION:
This study is a Randomized Clinical Trial, with individuals with morbid obesity, and will be consists of 3 groups:

1. Group 1 (G1 EXERCISE): This group will participate in an physical exercise program twice a week in hospital.
2. Group 2 (G2 - LIFESTYLE AND EXERCISE): This groups will receive the same G1 intervention associated with a weekly group followed up with techniques of cognitive behavioral therapy with a psychologist
3. Group 3 (G3 - CONTROL): This group will keep medical appointments information and routine procedure in the hospital.

Will be included in study the individuals with morbid obesity who do not have contraindications to practice low-intensity exercise.

Exclusion criteria are contraindications to physical exercise, individuals with cardiovascular disease with reduced functional capacity (class III and IV of the New York Heart Association), orthopedic problems, severe retinopathy, severe neuropathy, drug addicts and severe mental illness, metabolic or blood pressure decompensated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with morbid obesity
* Individuals do not have contraindications to practice low-intensity exercise.

Exclusion Criteria:

* Contraindications to physical exercise
* Cardiovascular disease with reduced functional capacity (class III and IV of the New York Heart Association)
* Orthopedic problems
* Severe retinopathy
* Severe neuropathy
* Drug addicts and severe mental illness
* High blood pressure or metabolic decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-11 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in Weight Loss | baseline and Four months

SECONDARY OUTCOMES:
Metabolic Parameters (composite) | baseline and Four months
  Metabolic parameters will be evaluated using total cholesterol, HDL, triglycerides and glucose (Assessment at baseline and 4 months).
Six minute walk test (6MWT) | baseline and Four months
  Functional capacity will be evaluated using the six minute walk test (6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Manoel R Trindade, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marcon ER, Gus I, Neumann CR. [Impact of a minimum program of supervised exercises in the cardiometabolic risk in patients with morbid obesity]. Arq Bras Endocrinol Metabol. 2011 Jun;55(5):331-8. doi: 10.1590/s0004-27302011000500006. Portuguese. PMID 21881816
- [Background] Fonseca Jr SJ, et al. Exercício Físico e Obesidade Mórbida: Uma Revisão Sistemática. ABCD Arq Bras Cir Dig 2013;26(Suplemento 1):67-73